CLINICAL TRIAL: NCT01115439
Title: Efficacy and Safety of Artesunate+Sulfadoxine-Pyrimethamine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Malaria Control Centers in Nangarhar, Kunar, Thakhar and Faryab Provinces of Afghanistan
Brief Title: Artesunate+Sulfadoxine-Pyrimethamine for the Treatment of Uncomplicated Falciparum Malaria
Acronym: ASPF
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: National Malaria and Leishmaniasis Control Program, Afghanistan (Other Government); World Health Organization (Other)
Responsible Party: Sponsor
Other Study IDs: BAKMAL1002
Record Dates: First submitted 2010-03-29; First posted 2010-05-04 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Falciparum Malaria
Keywords: falciparum malaria; artemisinin combination treatments
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- falciparum malaria: Febrile children (above six months of age) and non-pregnant adults with confirmed uncomplicated P. falciparum infection
  Interventions: Drug: artesunate plus sulfadoxine-pyrimethamine (AS+SP)

INTERVENTIONS:
Drug: artesunate plus sulfadoxine-pyrimethamine (AS+SP) — artesunate plus sulfadoxine-pyrimethamine (AS+SP)

SUMMARY:
In Afghanistan, studies over the past 15 years have shown a high degree of Plasmodium falciparum resistance to chloroquine (80%) and more recently an increasing degree of resistance to sulfadoxine-pyrimethamine monotherapy (12%). In 2003 the high failure rate of chloroquine against falciparum malaria led the national malaria treatment programme to switch its recommended first line drug treatment for uncomplicated Plasmodium falciparum malaria to artemisinin-based combination therapy (ACT) in the form of Artesunate/Sulfadoxine-Pyrimethamine (AS+SP). Second line drug treatment is oral quinine (7 days). The aim of this study is to conduct ongoing monitoring of the efficacy of the new combination against P. falciparum in a group of sentinel sites in Afghanistan.

DETAILED DESCRIPTION:
The objective of the study is to assess the efficacy and safety of Artesunate/Sulfadoxine-Pyrimethamine (AS+SP) for the treatment of uncomplicated P. falciparum infections in Nangarhar, Kunar, Thakhar, Faryab malaria control centers in Afghanistan.

This is an observational study. Patients will receive the recommended treatment for P. falciparum malaria in Afghanistan (Nangarhar, Kunar, Thakhar, Faryab malaria control centers). The participants will be febrile children above six months of age and non-pregnant adults with confirmed uncomplicated P. falciparum infection. Patients will be treated with AS+SP according to standard dosing regimens. Clinical and parasitological parameters will be monitored over a 42-day follow-up period to evaluate drug efficacy. The study will be conducted during the transmission season of falciparum malaria, i.e. October 2009 to January 2010 and September-December, 2010. Patients will be assessed clinically and via laboratory tests, particularly focussing on whether recurrences are recrudescences of the original infection or reinfections. All bio-medical findings will be recorded in specific patient case record forms and the electronic form of analyzed data as well as a final report will be sent to WHO-Afghanistan and National malaria control program offices for further actions. The patients will receive reasonable transportation costs for follow-up visits as well as one insecticide treated bed-net at the end of enrolment. The results of this study will be used to assist the Ministry of Health of Afghanistan in assessing the current national treatment guidelines for uncomplicated P. falciparum malaria.

ELIGIBILITY:
Inclusion:

* Age over six months.
* Mono-infection with P. falciparum detected by microscopy at a level of 500-150,000/µL asexual forms
* Presence of axillary or tympanic temperature ≥ 37.5 °C or oral or rectal temperature of ≥ 38 °C or history of fever during the past 24 h;
* ability to swallow oral medication;
* ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule; and
* Informed consent from the patient or from a parent or guardian in the case of children under 18 years of age.

Exclusion criteria:

* Presence of general danger signs in children aged under 5 years or signs of severe falciparum malaria according to the definitions of the World Health Organization (WHO)
* Mixed or mono-infection with another Plasmodium species detected by microscopy
* Presence of severe malnutrition (defined as a child whose growth standard is below -3 z-score, has symmetrical oedema involving at least the feet or has a mid-upper arm circumference < 110 mm)
* Presence of febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases, HIV/AIDS);
* Regular medication, which may interfere with antimalarial pharmacokinetics;
* History of hypersensitivity reactions or contraindications to any of the study medications;
* Female over 12 years of age

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Febrile children (above six months of age) and non-pregnant adults with confirmed uncomplicated P. falciparum infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-03; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients experiencing therapeutic failure | 42 days
  Proportion of patients experiencing therapeutic failure

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rahim Awab, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (4):
- Afghanistan (4):
  - Provincial Malaria Control Centers (MRC), Maymana, Faryab Province
  - Provincial Malaria Control Centers (MRC), Asadābād, Kunar
  - Provincial Malaria Control Centers (MRC), Jalalabad, Nangarhar
  - Provincial Malaria Control Centers (MRC), Taloqan

REFERENCES:
- [Derived] Awab GR, Imwong M, Pukrittayakamee S, Alim F, Hanpithakpong W, Tarning J, Dondorp AM, Day NP, White NJ, Woodrow CJ. Clinical trials of artesunate plus sulfadoxine-pyrimethamine for Plasmodium falciparum malaria in Afghanistan: maintained efficacy a decade after introduction. Malar J. 2016 Feb 25;15:121. doi: 10.1186/s12936-016-1167-z. PMID 26917051